CLINICAL TRIAL: NCT06742528
Title: Comparison Of Efficacy Of Iron Polymaltose Complex And Ferrous Sulphate In Iron Deficiency Anemia In Pediatric Patients With Iron Deficiency Anemia
Brief Title: Comparison Of Efficacy Of Iron Polymaltose Complex And Ferrous Sulphate In Iron Deficiency Anemia In Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arooj Khan (Other)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Sponsor-Investigator, Arooj Khan, Post Graduate Resident, Department of Child Health, Khyber Teaching Hospital
Organization: Khyber Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 591/DME/KMC
Record Dates: First submitted 2024-12-02; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Iron Deficiency Anemia; Iron Deficiency, Anaemia in Children
Keywords: IRON POLMALTOSE COMPLEX; FERROUS SULPHATE; Iron Deficiency, Anaemia in Children
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferrous sulfate; teferrol

STUDY DESIGN:
Intervention Model Description: Brief history and demographic data including age, gender, duration of pallor, residence, weight, educational level of mother, socioeconomic status of father will be noted. Under aseptic techniques 5cc venous sample will be drawn and send to hospital laboratory for baseline hemoglobin and serum ferritin level. All patients will be dewormed before starting therapy by giving oral albendazole l0 ml stat dose. Patients will be divided randomly in two groups using blocked randomization generated by computer software. Group A will be given ferrous sulphate in a dose of 6mg/kg/day of elemental iron once daily for 8 weeks orally in syrup form. Group B will be given Iron Polymaltose complex in a dose of 6mg/kg/day of elemental iron once daily orally for 8 weeks. Both the groups will be called for follow up. Hemoglobin level will be assessed after 8 week of therapy.
Who Masked: Participant
Masking Description: Patients will be divided randomly in two groups using blocked randomization generated by computer software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Ferrous sulphate) (Active Comparator): Group A will be given Ferrous sulphate in a dose of 6mg/kg/day of elemental iron once daily for 8 weeks orally in syrup form.
  Interventions: Drug: Ferrous sulfate
- Group B (Iron Polymaltose complex) (Active Comparator): Group B will be given Iron Polymaltose complex in a dose of 6mg/kg/day of elemental iron once daily orally for 8 weeks.
  Interventions: Drug: Iron Polymaltose Complex

INTERVENTIONS:
Drug: Ferrous sulfate — ferrous sulphate in a dose of 6mg/kg/day of elemental iron once daily for 8 weeks orally in syrup form.
  Arms: Group A (Ferrous sulphate)
Drug: Iron Polymaltose Complex — Iron Polymaltose complex in a dose of 6mg/kg/day of elemental iron once daily orally for 8 weeks.
  Arms: Group B (Iron Polymaltose complex)

SUMMARY:
This study aims to compare the efficacy of two iron preparation for the management of children presented with iron deficiency anemia. Ferrous sulphate and lron polymaltose (ferric form) are most commonly used preparations. Both drugs are easily available in market and are often recommended by pediatriclans. The efficacy, bioavail.tbilily, side effects and cost of these preparations vary. This study is designed to find out a drug with better efficacy that can be used for treatment of iron deficiency anemia in local population.

DETAILED DESCRIPTION:
Anemia remains a condition with high prevalence in populations worldwide. It is predominantly associated with nutritional status and socioeconomic conditions or hereditary diseases. The majority of anemia cases are linked to iron deficiency-named iron-deficiency anemia resulting from low intake of iron-rich foods in the diet, or from substantial blood loss.

This study aims to compare the efficacy of two iron preparation for the management of children presented with iron deficiency anemia. Ferrous sulphate and lron polymaltose (ferric form) are most commonly used preparations. Both drugs are easily available in market and are often recommended by pediatriclans. The efficacy, bioavail.tbilily, side effects and cost of these preparations vary. This study is designed to find out a drug with better efficacy that can be used for treatment of iron deficiency anemia in local population.

ELIGIBILITY:
Inclusion Criteria:

* Patients having iron deficiency anemia

Exclusion Criteria:

1. Patients diagnosed as congenital aplastic anemia or thalassemia (Determined from medical record).
2. Patients who were transfused in previous 4 weeks (will be determined on history)
3. Children having mal-absorption syndrome and diarrheal illnesses. (will be determined on history and medical record)
4. Gastrointestinal bleeding suggested by history of hematemesis (bloody vomit), melena (black colored stools) or bloody stools.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Increase Of Hemoglobin Level | 8 weeks
  Increase in Hemoglobin level measured by a Complete Blood Count as compared to pre treatment Hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montoro-Huguet MA, Santolaria-Piedrafita S, Canamares-Orbis P, Garcia-Erce JA. Iron Deficiency in Celiac Disease: Prevalence, Health Impact, and Clinical Management. Nutrients. 2021 Sep 28;13(10):3437. doi: 10.3390/nu13103437. PMID 34684433
- [Background] Martin-Masot R, Nestares MT, Diaz-Castro J, Lopez-Aliaga I, Alferez MJM, Moreno-Fernandez J, Maldonado J. Multifactorial Etiology of Anemia in Celiac Disease and Effect of Gluten-Free Diet: A Comprehensive Review. Nutrients. 2019 Oct 23;11(11):2557. doi: 10.3390/nu11112557. PMID 31652803
- [Background] Rockey DC, Altayar O, Falck-Ytter Y, Kalmaz D. AGA Technical Review on Gastrointestinal Evaluation of Iron Deficiency Anemia. Gastroenterology. 2020 Sep;159(3):1097-1119. doi: 10.1053/j.gastro.2020.06.045. Epub 2020 Aug 21. No abstract available. PMID 32828801
- [Background] Zheng J, Liu J, Yang W. Association of Iron-Deficiency Anemia and Non-Iron-Deficiency Anemia with Neurobehavioral Development in Children Aged 6-24 Months. Nutrients. 2021 Sep 28;13(10):3423. doi: 10.3390/nu13103423. PMID 34684422
- [Background] Orsango AZ, Habtu W, Lejisa T, Loha E, Lindtjorn B, Engebretsen IMS. Iron deficiency anemia among children aged 2-5 years in southern Ethiopia: a community-based cross-sectional study. PeerJ. 2021 Jun 28;9:e11649. doi: 10.7717/peerj.11649. eCollection 2021. PMID 34249504
- [Result] Paulino CTDS, Nishijima M, Sarti FM. Association of Iron Supplementation Programs with Iron-Deficiency Anemia Outcomes among Children in Brazil. Nutrients. 2021 Apr 30;13(5):1524. doi: 10.3390/nu13051524. PMID 33946398